CLINICAL TRIAL: NCT05226299
Title: Cough Desensitization Therapy for Cough Hypersensitivity Syndrome: Pilot 2
Brief Title: Cough Desensitization Therapy: Pilot 2
Acronym: CDTPilot2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Montana (Other)
Responsible Party: Principal Investigator, Laurie Slovarp, Professor, University of Montana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UMontana
Record Dates: First submitted 2022-01-25; First posted 2022-02-07 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Cough
Keywords: chronic cough; refractory chronic cough; cough hypersensitivity
MeSH Terms: conditions — Cough; Chronic Cough | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: One group will receive the placebo treatment while the second group receives the active treatment.
Who Masked: Participant
Masking Description: Participants will be blinded to group assignment (active treatment vs. placebo).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental: Supra-threshold capsaicin (Experimental): Arm: Experimental: Supra-threshold capsaicin Participants will be exposed to progressively increasing concentrations of aerosolized capsaicin (the ingredient in chili peppers that makes them spicy, and a known cough stimulant) to stimulate an urge-to-cough. Participants will be coached to implement cough suppression strategies following each exposure.
  Interventions: Biological: Supra-threshold and progressive doses of diluted capsaicin via a dosimeter-controlled nebulizer
- Arm: Placebo Comparator: Saline (Placebo Comparator): Participants will be exposed repeatedly to aerosolized saline through a nebulizer during treatment.
  Interventions: Biological: Saline

INTERVENTIONS:
Biological: Supra-threshold and progressive doses of diluted capsaicin via a dosimeter-controlled nebulizer — Participants will be exposured to increasing doses of aerosolized capsaicin (a known cough stimulant) through a dosimeter-controlled nebulizer, while implementing behavioral cough suppression strategies. The concentration of capsaicin will increase incrementally as tolerated, as long as participants are still able to suppress cough. Individual doses will never exceed 1000 micromolar. Cumulative doses per session will never exceed 2000 micromolar. Participants will attend 12 treatment sessions and be given up to 12 exposures per treatment session. Participants will be encouraged to use cough suppression strategies outside of treatment sessions as much as possible to attempt to suppress cough.
  Arms: Experimental: Supra-threshold capsaicin
Biological: Saline — Participants will be repeatedly exposed to a saline through a dosimeter-controlled nebulizer during treatment sessions. Participants will attend 12 treatment sessions and be given up to 12 exposures per treatment session.
  Arms: Arm: Placebo Comparator: Saline

SUMMARY:
The purpose of this study is to investigate a modified behavioral treatment for chronic cough due to cough hypersensitivity syndrome (CHS). This type of CC is a non-productive cough that is due, in part, to over-expression of transient receptor potential vanilliod (TRPV) receptors in the airway epithelium, which contribute to a dry cough elicited by typically non-tussive stimuli (e.g., cold air, smells) or by low doses of tussive stimuli (e.g., smoke). Currently available treatment options are limited to neuromodulator medications (e.g., gabapentin, amytriptiline) and behavioral cough suppression therapy (BCST), neither of which is 100% effective. The primary component of BCST is teaching patients to suppress their cough in the presence of an urge-to-cough. Studies have confirmed a reduction in cough sensitivity (as tested with inhaled capsaicin) following 1-4 weeks of successful cough suppression. However, patients with severe CHS are not able to suppress their cough in the presence of uncontrollable environmental stimuli and, hence, do not respond well to the therapy. The purpose of this study is to determine the potential of treating CHS by implementing BCST while stimulating cough with progressive concentrations of inhaled diluted aerosolized capsaicin. The investigators hypothesize this treatment will result in a reduction in cough-reflex sensitivity, cough-related quality of life, and cough frequency.

DETAILED DESCRIPTION:
The study will be a randomized, placebo-controlled, blinded study. It will take place in three phases, across 10 weeks.

WEEK 1: BASELINE TESTING AND TRAINING (approximate time = 1 hour).

Cough sensitivity testing: Standardized procedures that have been established and approved by the FDA will be used to determine cough sensitivity. Participants will inhale capsaicin vapor (a known cough stimulant) through a nebulizer with dosimeter, that delivers a specific dose of capsaicin in a mist form. They will inhale doubling doses of capsaicin mist from .49 micromolar to 1000 micromolar. The testing will be stopped when the investigators find the dose that causes five coughs or after giving the 1000 micromolar dose, whichever comes first. This testing will take approximately 30 minutes.

Urge-to-cough (UTC) testing: Participants be asked to report their UTC on a scale from 0 (no UTC) to 10 (maximum UTC) after each mist of capsaicin and after being presented with the following stimulants/tasks that cause some people to cough: perfume, bleach, vinegar, wood chips, laundry soap, cleaning wipe, deep and fast breath through the mouth, sustained voicing, reading a 55 word passage, and yelling a short phrase). This testing will take about 10 minutes.

Cough-related quality of life: Participants will complete the Leicester Cough Questionnaire which is a 23-item validated questionnaire designed to measure cough-related quality of life. It will take about 5 minutes.

Visual analogue cough severity (VAS): Participants will rate their cough severity on a visual analogue scale by placing a tick mark on a 100 mm line where 0 mm indicates "no cough" and 100 mm indicates "worst possible cough".

WEEKS 2-7: TREATMENT. Participants will attend treatment sessions twice per week for up to six weeks. Participants will use the breathing strategies following inhalation of either the active substance (experimental condition) or repeated exposures to an inactive substance (placebo condition). Participants will do this no more than twelve times per session. Each session will take 45-60 minutes. If a participant misses a treatment session, the investigators will attempt to re-schedule that session. Each participant must complete at least 10 treatment sessions to remain in the study.

WEEKS 8 AND 10: POST-TREATMENT TESTING. Outcome measures, as in the baseline phase, will be taken at one-week and three-weeks post-treatment. The LCQ will be measured again at three-months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Currently suffering from a cough that started at least 8 weeks ago
* Have seen at least one physician for the cough and have received medical treatment without success
* Normal chest x-ray, pulmonary function testing (completed by your physician or a qualified speech-language pathologist).
* Completion of a laryngoscopy (by ENT physician or qualified speech-language pathologist) with no evidence of an anatomical abnormality (i.e., masses or lesions such as nodules, cysts, or cancer) that could contribute to cough.
* Willing to take a pregnancy test before enrollment (if applicable)
* Willing to use contraception during the study (if applicable; we will not be able to supply you with contraceptive methods)
* If you are diagnosed with asthma, you may enroll in the study if you are regularly followed by a pulmonologist who will verify, in writing, that your asthma symptoms are well-controlled (apart from cough symptoms) with your current medication protocol, which would not be altered when you are in the study. In order to remain in the study, your forced expiratory volume (FEV1), which will be measured during baseline lung function testing with spirometry, must be no less than 60% of predicted values given age, height, and weight. You must also carry a rescue inhaler with you when participating in all assessment and treatment sessions.
* Willing to sign an informed consent form

Exclusion Criteria:

* Under 18 years of age
* Positive for COVID-19 or presenting with any of the following symptoms of COVID- 19: fever or chills, sputum, difficulty breathing, fatigue, muscle or body aches, headache, loss of taste or smell, sore throat, congestion or runny nose, nausea or vomiting, diarrhea.
* Have not followed current local, state, and CDC COVID-19 mitigation guidance, especially regarding travel.
* Unwilling to comply with COVID-19 precautions (see below)
* Currently a smoker of any substance
* Pregnant or attempting to become pregnant
* Diagnosed with a respiratory or pulmonary condition (other than asthma) that commonly contributes to cough (e.g., chronic obstructive pulmonary disease, emphysema, lung cancer, bronchitis)
* Diagnosed with asthma that is not well managed and/or do not have the necessary written consent by a pulmonologist to be in the study.
* Suffering from any signs of upper respiratory illness
* Taken any of the following medications within the past month:

  * lisinopril/Prinivil/Zestril
  * captopril/Capoten
  * enalapril/Epaned/Asotec, ramipril/Altace
  * benazepril/Lotensin
  * fosinopril/Monopril
  * moexipril/Univasc
  * perindopril/Aceon
  * quinapril/Accupril
  * trandolapril/Mavik

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline Leicester Cough Questionnaire (LCQ) score at 1 week post-treatment | The LCQ will be measured before treatment (baseline) and 1 week post treatment
  The LCQ is a 23-item validated patient-report questionnaire that takes about 5 minutes to fill out. It results in three domain scores (Social, Psychological, and Physical) and one Total score, which is the sum of the domain scores. Domain scores are between 1 and 7. The total score is between 3 and 21. A higher score means a better outcome.
Change from baseline visual analogue cough severity score at 1 week post-treatment | Cough severity will be will be measured before treatment (baseline) and 1 week post-treatment
  Participant's perceived cough severity will be measured using a visual analogue scale. They will place a tick mark on a 100 mm line where 0mm indicates "no cough problem" and 100 mm indicates "worst possible cough problem".

SECONDARY OUTCOMES:
Change from baseline cough-reflex sensitivity at 1 week post-treatment | Cough-reflex sensitivity will be measured before treatment (baseline), and 1 week post-treatment
  Cough sensitivity will be measured with cough challenge testing. Standardized procedures that have been established and approved by the FDA will be used. Participants will inhale capsaicin vapor (a known cough stimulant) through a nebulizer with dosimeter, that delivers a specific dose of capsaicin in a mist form. They will inhale doubling doses of capsaicin mist from .49 micromolar to 1000 micromolar. The testing will be stopped when the investigators find the dose that causes five coughs or after giving the 1000 micromolar dose, whichever comes first. This testing will take approximately 30 minutes.
Change from baseline urge-to-cough (UTC) testing at 1 week post-treatment | UTC testing will be measured before treatment (baseline) and 1 week post-treatment
  During UTC testing, participants will be asked to report their perceived UTC on a scale from 0 (no UTC) to 10 (maximum UTC) after each exposure to capsaicin during cough-reflex sensitivity testing as well as after being presented with the following stimulants/tasks that cause some people to cough: perfume, bleach, laundry soap, fabric softener, vinegar, scented candle, deep and fast breath through the mouth twice in a row, sustained voicing, reading a 55 word passage, and yelling a short phrase. This testing will take about 10 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Slovarp, PhD, Principal Investigator — University of Montana
Locations (1):
- University of Montana, Missoula, Montana, United States

REFERENCES:
- [Derived] Slovarp LJ, Reynolds JE, Tolbert S, Campbell S, Welby S, Morkrid P. Cough desensitization treatment for patients with refractory chronic cough: results of a second pilot randomized control trial. BMC Pulm Med. 2023 Apr 28;23(1):148. doi: 10.1186/s12890-023-02423-6. PMID 37118696